CLINICAL TRIAL: NCT03163927
Title: The Effect of Simulation-Based Training on Performance and Stress in the Clinical Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Mikael Johannes Vuokko Henriksen, Principal Investigator, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: StressLBP
Record Dates: First submitted 2017-04-24; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Spinal Puncture Complications; Simulation-based Training; Stress, Emotional
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive a 1.5-hour standardized simulation-based training course, with mastery learning.
  Interventions: Other: Simulation-based training
- Control (No Intervention): Participants observe a procedure performed by a senior.

INTERVENTIONS:
Other: Simulation-based training — See arm description
  Arms: Intervention

SUMMARY:
This study will investigate the effect of simulation-based training with mastery learning (SBML) on novice performers' lumbar puncture (LP) performance in a clinical setting. The study will investigate the effect on operators' performance, stress level, and on patient experienced stress, confidence in operator, and patient-related outcomes of pain, and risk of subsequent Post Dural Puncture Headache (PDPH), and days of sickness leave.

The study will compare the effect of the training to a control group of novices receiving standard training and additionally to an intermediate and an expert group.

The study will provide insight into the translational effect from the simulation based setting to clinical performance. Further, the study will explore: if stress decreases operators' performance; if operators stress affects the patient stress level; and the effect of SBML on patient-related outcomes.

DETAILED DESCRIPTION:
The lumbar puncture procedure is considered a complex procedure. Junior doctors hold uncertainties in performing the procedure and perform below stakeholders expectations. This conflicts with the potential need for immediate performance on critical patients.

The traditional training for junior physicians has been guided by the expectation that experience will lead to mastery. This assumption has been disproved by simulation based and observational studies calling for more educational research including its impact on patient outcomes. A contrast to the maxim of "see one, do one, teach one" is mastery learning (ML). ML implies that learners should practice and re-test until they reach a designated mastery level, making the final level the same for all, although the time taken to reach that level may vary.

Novices trained by simulation based training with mastery learning (SBML) achieve a higher performance level than more experienced physicians only having received clinical training. However, the translational effect into the clinical context is unknown as the training and assessment of competence was performed in the simulation based setting, not integrating aspects as patient communication and positioning. For the lumbar puncture, the complexity of the procedure pertains to both technical and non-technical aspects as patient interaction, communication, the corporation with the assistant and environmental conditions.

Hence, there is a need for more knowledge on the effect of simulation-based training with mastery learning for junior doctors' performance in the clinical setting which should include the effect on patient-related outcomes.

As novices describe a fear of doing harm and hold performance related uncertainty, they may be susceptible to experience a stress sensation. Stress during performance of clinical procedures reduces the working memory and is associated with impaired performance. Expert performers' reports that stress during the procedure performance might be transmitted to the patient. Patients experiencing stress during the procedure holds a significantly increased risk of a prolonged duration of post dural puncture headache.

Stress- stimuli, experience, and responses are complex, as the judgment on whether a situation is perceived as pleasant or threatening depends on the individuals' appraisal, which is based: on previous experience; previous learning; the setting and expectations of the outcome. Stress stimuli arise when the appreciation of the situation is negative. Performers holding a strategy for their performance during stress are less prone to experience a stress sensation. Hence, the integration of a strategy for performing the procedure, based on the experts' process goals might benefit novices' risk of experiencing stress during procedure performance. The effect on such stress reduction to the patient experience of stress and the risks of procedure-related side effects has never been investigated.

The aim of this study is to investigate the effect of simulation-based training with mastery learning on novices' lumbar puncture performance, patient related outcomes and stress experienced by the physicians and patients during the procedure. The effect and outcomes will be compared with intermediate and expert lumbar puncture performers.

ELIGIBILITY:
For the medical doctors randomized:

Inclusion Criteria:

* MD, or Medical student working as substitute junior medical officer, or having clinical rotation at the study sites.
* Speaking Danish fluently

Exclusion Criteria:

* Previous Lumbar Puncture experience
* Previous formal training in the lumbar puncture procedure

Eligible patients:

Inclusion criteria:

* Glasgow Coma Scale 15
* Referred to the outpatient clinic for a lumbar puncture.
* Proficiency in the Danish Language
* Age between 18 and 80 years
* Understand study implications and co-operate without a need for personal assistance.
* Providing written and orally informed consent

Exclusion criteria for patients:

* Lumbar puncture intended on suspicion of Alzheimer or other dementia diagnosis.
* Cognitive impairment, assessed by the study investigator or local nurse/doctor
* Physical disabilities, requiring personal assistance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Performance | Videos will be recorded at time of lumbar puncture performance, for subsequent ratings within 3 months.
  Performance of the procedure assessed by the Lumbar Puncture Assessment Tool (LumPAT)
Doctors Heart Rate Variability before performance (Heart rate) | A recording of 5 minutes obtainted five minutes before performance, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: Heart rate (bp/min);
Doctors Heart Rate Variability before performance (Power) | A recording of 5 minutes obtainted five minutes before performance, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: Power of Low Frequency, Very Low frequency, High Frequency (ms), a ratio of LF/HF will be calculated
Doctors Heart Rate Variability before performance | A recording of 5 minutes obtainted five minutes before performance, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: RMSDD (ms)
Doctors Heart Rate Variability before performance (pNN50) | A recording of 5 minutes obtainted five minutes before performance, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: pNN50 (%)
Doctors Heart Rate Variability during performance (Heart rate) | A recording of 5 minutes obtainted five minutes before obtaining liquor, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: Heart rate (bp/min);
Doctors Heart Rate Variability during performance (Power) | A recording of 5 minutes obtainted five minutes before obtaining liquor, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: Power of Low Frequency, Very Low frequency, High Frequency (ms), a ratio of LF/HF will be calculated
Doctors Heart Rate Variability during performance (RMSDD) | A recording of 5 minutes obtainted five minutes before obtaining liquor, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: RMSDD (ms)
Doctors Heart Rate Variability during performance (pNN50) | A recording of 5 minutes obtainted five minutes before obtaining liquor, is compared to a rest-state recording after the procedure performance
  Heart Rate Variability: pNN50 (%)
Doctors State Trait Anxiety Inventory - Short | Five minutes before performance; Just Before Needle insertion;
  A questionaire exploring the stress related anxiety (scores range from 6-24)
Doctors Cognitive Appraisal | Five minutes before performance
  Cognitive Appraisal explores the individuals perception of resources and demands for the performance (scores range from 1/6 to 6)

SECONDARY OUTCOMES:
Patient Heart Rate Variability before performance | A recording of 5 minutes obtained five minutes before performance
  Heart Rate Variability: Heart rate (bp/min);
Patient Heart Rate Variability during performance | A 5 minutes recording during procedure handling, just before obtaining liquor.
  Heart Rate Variability: Heart rate (bp/min);
Patient Heart Rate Variability before performance | A recording of 5 minutes obtained five minutes before performance
  Heart Rate Variability: Power of Low Frequency, Very Low frequency, High Frequency (ms), a ratio of LF/HF will be calculated
Patient Heart Rate Variability during performance | A 5 minutes recording during procedure handling, just before obtaining liquor.
  Heart Rate Variability: Power of Low Frequency, Very Low frequency, High Frequency (ms), a ratio of LF/HF will be calculated
Patient Heart Rate Variability before performance | A recording of 5 minutes obtained five minutes before performance
  Heart Rate Variability: RMSDD (ms)
Patient Heart Rate Variability during performance | A 5 minutes recording during procedure handling, just before obtaining liquor.
  Heart Rate Variability: RMSDD (ms)
Patient Heart Rate Variability before performance | A recording of 5 minutes obtained five minutes before performance
  Heart Rate Variability: pNN50 (%)
Patient Heart Rate Variability during performance | A 5 minutes recording during procedure handling, just before obtaining liquor.
  Heart Rate Variability: pNN50 (%)
Patients State Trait Anxiety Inventory - Short | Five minutes before performance; Just Before Needle insertion; Five minutes after termination of the procedure
  A questionaire exploring the stress related anxiety (scores range from 6-24)
Procedure outcomes | Registrered during procedure operation
  Number of needle insertions, Failing/abandoning the procedure performance (yes/no)
Duration of time to needle insertion | Registrered during procedure operation, or evaluated using the videorecordings of the procedure
  Time from needle penetration of the skin to obtaining liquor (mm:ss)
Confidence in operator | Five minutes after termination of the procedure
  A 10-point Likert scale: 0=not confident - 10=very confident
Pain intensity during procedure | Five minutes after termination of the procedure
  A 10-point Likert scale; 0= no pain - 10= Worst imaginable pain.
Post Dural Puncture Headache | Telephone interview seven days after the procedure performance date
  Post Dural Puncture Headache, using the Lübeckers classification
Days of sickness leave | Telephone interview seven days after the procedure performance date
  Days sick leave related to procedure performance

CONTACTS AND LOCATIONS:
Overall Officials: Mikael J Henriksen, MD, Principal Investigator — CAMES - Rigshospitalet
Locations (3):
- Denmark (3):
  - Department of Neurology, Rigshospitalet - Glostrup, Glostrup Municipality, Capital Region of Denmark
  - Department of Neuology, Herlev Hospital, Herlev, Capital Region of Denmark
  - Department of Neurology, University Hospital Zealand, Roskilde, Region Sjælland

IPD SHARING:
Plan to Share IPD: No